CLINICAL TRIAL: NCT02634242
Title: Study on the Antiaging Effect of Chinese Herb Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Chin Kun Wang, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: CS08008
Record Dates: First submitted 2015-12-08; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Gynecological Disorders
Keywords: Si Wu Tang; antioxidation; anthropometric measurements; liver; skin
MeSH Terms: conditions — Genital Diseases, Female | interventions — si-wu-tang

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Si-Wu-Tang (SWT) (Experimental): Subjects are recommended to drink 125 mL of SWT (n=30) for 6 continuous days per month during the following 6 months and vice versa with one month of washout period in between.
  Interventions: Other: Si-Wu-Tang (SWT); Other: placebo
- placebo (Placebo Comparator): Subjects are recommended to drink 125 mL of Placebo (n=30) for 6 continuous days per month during the following 6 months and vice versa with one month of washout period in between.
  Interventions: Other: Si-Wu-Tang (SWT); Other: placebo

INTERVENTIONS:
Other: Si-Wu-Tang (SWT) — The purpose of the current study was to check the physiological improvement of SWT on liver and skin and also the antioxidation in healthy adults.
  Other Names: Si-Wu-Tang (SWT) is a Traditional Chinese Medicine formula
Other: placebo — The purpose of the current study was to check the physiological improvement of placebo on liver and skin and also the antioxidation in healthy adults.

SUMMARY:
The purpose of the current study was to check the physiological improvement of SWT on liver and skin and also the antioxidation in healthy adults.

DETAILED DESCRIPTION:
Background: Si-Wu-Tang (SWT) is a well-known traditional Chinese medicine (TCM) and widely used for treating various gynecological disorders. The purpose of the current study was to check the physiological improvement of SWT on liver and skin and also the antioxidation in healthy adults.

Methods: Sixty healthy voluntary subjects were recruited and assigned into two groups, who drank 125 mL of placebo (n=30) or SWT (n=30) for 6 continuous days per month during the following 6 months and vice versa with one month of washout period in between. During the initial, 3rd, 6th, 10th, and 13th months anthropometric measurements were performed as well as fasting blood samples were drawn for various biochemical assays. Abdominal ultrasonic and skin examination were performed at the initial, 6th and 13th months.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* exclusion criteria were history of smoking, alcoholism
* pregnant or lactating women,
* chronic diseases, hepatic or renal dysfunction.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Total thiobarbituric acid reactive substances (TBARS) | 6 months

SECONDARY OUTCOMES:
Glutathione content (GSH) | 6 months
Total antioxidant capacity (TEAC)activities. | 6 months
Superoxide dismutase (SOD) activity | 6 months
GPx and glutathione reductase (GR) activity | 6 months
Catalase | 6 months
Glutamic oxaloacetic transaminase (GOT) | 6 months
Glutamic pyruvic transaminase (GPT) | 6 months

OTHER OUTCOMES:
Skin sebum content | 6 months
Skin hydration | 6 months
Skin surface water loss | 6 months
Skin melanin index | 6 months
Skin elasticity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Kun Wang, Study Chair — Chung Shan Medical University